CLINICAL TRIAL: NCT00007930
Title: Randomized Trial of Wide Mesorectal Excision Versus Total Mesorectal Excision for Mid Rectal Cancer
Brief Title: Comparison of Two Types of Surgery in Treating Patients With Rectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Medical Research Council (NMRC), Singapore (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068354; NMRC-ICR01; EU-99019
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2006-12

CONDITIONS: Colorectal Cancer
Keywords: stage I rectal cancer; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Laparoscopy

INTERVENTIONS:
Procedure: conventional surgery
Procedure: laparoscopic surgery

SUMMARY:
RATIONALE: Surgery to remove the tumor may be an effective treatment for rectal cancer. It is not yet known whether one type of surgery is more effective than another for rectal cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two types of surgery in treating patients who have rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare local and distant recurrences in patients with mid-rectal cancer treated with wide mesorectal surgical excision with straight colorectal anastomosis versus total mesorectal surgical excision with colonic J pouch coloanal anastomosis.
* Compare the functional, physiological, and anatomical outcomes in these patients treated with these two surgical procedures.
* Compare disease-free survival and overall survival in these patients treated with these two surgical procedures.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to treatment center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo surgical resection with a wide mesorectal excision followed by a straight colorectal anastomosis.
* Arm II: Patients undergo surgical resection with a total mesorectal excision followed by a colonic J pouch coloanal anastomosis. Patients then receive a temporary ileostomy which is closed 6 weeks later.

Patients are followed at 6 weeks, every 4-6 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A minimum of 800 patients (400 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinical diagnosis of rectal cancer by colonoscopy or barium enema

  * Distal margin of tumor arises within 9-15 cm from the anal verge as measured by rigid sigmoidoscopy
* No synchronous multiple adenocarcinomas
* Candidate for low anterior surgical resection by laparoscopy or conventional open method
* No evidence of gross metastatic disease
* No evidence of peritoneal or pelvic metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* At least 6 months

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other malignancy within the past 5 years

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Neoadjuvant or adjuvant chemoradiotherapy allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* See Chemotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 1999-08

PRIMARY OUTCOMES:
Local recurrence at 3 years

SECONDARY OUTCOMES:
Disease-free and overall survival at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Heah Sieu Min, MD, Study Chair — National Cancer Centre, Singapore
Locations (3):
- China (2):
  - Hong Kong Sanatorium & Hospital, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
- National Cancer Centre - Singapore, Singapore, Singapore